CLINICAL TRIAL: NCT02543255
Title: Anti-Androgens and Cabazitaxel in Defining Complete Response in Prostatectomy (ACDC-RP Trial): A Randomized, Open-label, Multi-centre Phase-2 Study Evaluating the Pathological Complete Response (pCR) Rate Following Neoadjuvant Therapy in Participants With High-risk Prostate Carcinoma for Whom Radical Prostatectomy is Indicated
Brief Title: Anti-Androgens and Cabazitaxel in Defining Complete Response in Prostatectomy (ACDC Trial)
Acronym: ACDC-RP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-051
Record Dates: First submitted 2015-09-03; First posted 2015-09-07 (Estimated); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer
Keywords: High risk
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Prednisone; Leuprolide; cabazitaxel; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Abiraterone acetate + prednisone + leuprolide + cabazitaxel (Experimental): Participants randomized to this arm will receive abiraterone acetate (1000 mg/day), prednisone (5 mg twice daily), leuprolide (22.5 mg every 3 months), and cabazitaxel (20 mg/m2, with 6 mg pegfilgrastim administered 24 h following cabazitaxel) prior to radical prostatectomy.
  Interventions: Drug: Abiraterone acetate with prednisone; Drug: Leuprolide; Drug: Cabazitaxel with peg-filgrastim
- Abiraterone acetate + prednisone + leuprolide (Active Comparator): Participants randomized to this arm will receive abiraterone acetate (1000 mg/day) , prednisone (5 mg twice daily), and leuprolide (22.5 mg every 3 months) prior to radical prostatectomy.
  Interventions: Drug: Abiraterone acetate with prednisone; Drug: Leuprolide

INTERVENTIONS:
Drug: Abiraterone acetate with prednisone — Abiraterone acetate will be administered orally as a tablet at 1000 mg/day with prednisone (5 mg oral tablet, twice daily) for 24 weeks.
Drug: Leuprolide — Leuprolide will be administered by subcutaneous injection at 22.5 mg dose every 12 weeks for 24 weeks.
Drug: Cabazitaxel with peg-filgrastim — Cabazitaxel will be administered in 6 cycles, with 20 mg/m2 per cycle and 3 weeks between cycles.
  Arms: Abiraterone acetate + prednisone + leuprolide + cabazitaxel

SUMMARY:
This study evaluates the use of chemotherapy with cabazitaxel in addition to abiraterone acetate, prednisone, and leuprolide in neoadjuvant setting prior to radical prostatectomy in patients with high-risk prostate carcinoma. Half of the participants will receive treatment with abiraterone acetate, prednisone, leuprolide, and cabazitaxel, while the other half will receive only abiraterone acetate, prednisone, and leuprolide.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent;
* Histologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features with a minimum of 3 cores positive for tumour;
* Tumour biopsy tissue accessible for downstream evaluation;
* Must be candidates for radical prostatectomy and considered surgically resectable by urologic evaluation;
* High Risk D'Amico score defined as either PSA > 20, Gleason score ≥ 8 as determined by the local pathologist; or T2c-3 based on DRE, pathologic review +/- imaging;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1;
* No evidence of metastatic disease or nodal disease as determined by radionuclide bone scans and computed tomography (CT)/magnetic resonance imaging (MRI); non-pathological lymph nodes must be less than 15 mm in the short (transverse) axis;
* Able to swallow the study drug(s) as prescribed and comply with study requirements;
* Required initial laboratory values:
* Absolute neutrophil count (ANC) ≥ 1500/μL;
* Platelet count ≥ 100,000/μL;
* Hemoglobin ≥ 90 g/L;
* Creatinine ≤ 175 μmol/L;
* Bilirubin ≤ upper limit of institutional normal (ULN);
* AST/ALT ≤ 1.5 × ULN.

Exclusion Criteria:

* Received an investigational agent within 4 weeks prior to screening;
* Stage T4 prostate cancer by clinical examination or radiologic evaluation;
* Hypogonadism or severe androgen deficiency as defined by screening serum testosterone below the normal range for the institution;
* Prior androgen deprivation, chemotherapy, surgery, or radiation for prostate cancer;
* Receiving concurrent androgens, estrogens, or progestational agents, or received any of these agents within the 6 months prior to randomization;
* History of another malignancy within the previous 5 years other than curatively treated nonmelanomatous skin cancer and non-muscle invasive bladder cancer;
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, cardiovascular disease, unstable angina pectoris, cardiac arrhythmia that is symptomatic or requires active therapy; deep venous thrombosis within 3 months prior to randomization;
* Previous use, or participation in a clinical trial, of an investigational agent that blocks androgen synthesis (e.g., abiraterone acetate, TAK-700, TAK-683, TAK-448) or targets the androgen receptor (e.g., enzalutamide, BMS 641988);
* Liver injury or disease (e.g., viral hepatitis, liver failure Child-Pugh Class C).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Pathological complete response | 24 weeks from start of treatment.

SECONDARY OUTCOMES:
Pre-operative PSA levels | 24 weeks of treatment
  The effect of neoadjuvant leuprolide, and abiraterone acetate and prednisone with and without cabazitaxel on pre-operative PSA will be evaluated.
Mean nadir PSA levels | 24 weeks of treatment
  The effect of neoadjuvant leuprolide, abiraterone acetate, and prednisone with and without cabazitaxel on mean nadir PSA levels will be evaluated.
Percentage of participants achieving a PSA < 0.2 ng/mL | 24 weeks of treatment
  The percentage of participants achieving a PSA < 0.2 ng/mL following treatment with neoadjuvant leuprolide, abiraterone acetate, and prednisone with and without cabazitaxel will be evaluated.
Percentage of participants achieving a 50 and 90% decrease in PSA levels | up to 24 weeks of treatment
  The percentage of participants achieving a 50 and 90% decrease in PSA levels following treatment with neoadjuvant leuprolide, abiraterone acetate, and prednisone with and without cabazitaxel will be evaluated.
Rate of positive surgical margins | up to 24 weeks of treatment
  The rate of positive surgical margins following treatment with neoadjuvant leuprolide, abiraterone acetate, and prednisone with and without cabazitaxel will be evaluated.
Rate of near-complete response (<5 mm tumour) | up to 24 weeks of treatment
  The rate of near-complete response (<5 mm tumour) following treatment with neoadjuvant leuprolide, abiraterone acetate, and prednisone with and without cabazitaxel will be evaluated.
Rate of extracapsular extension | up to 24 weeks of treatment
  The rate of extracapsular extension following treatment with neoadjuvant leuprolide, abiraterone acetate, and prednisone with and without cabazitaxel will be evaluated.
Rate of positive seminal vesicle involvement | up to 24 weeks of treatment
  The rate of positive seminal vesicle involvement following treatment with neoadjuvant leuprolide, abiraterone acetate, and prednisone with and without cabazitaxel will be evaluated.
Rate of nodal involvement | up to 24 weeks of treatment
  The rate of nodal involvement following treatment with neoadjuvant leuprolide, abiraterone acetate, and prednisone with and without cabazitaxel will be evaluated.
Tumour proliferation (Ki-67 index) | up to 24 weeks of treatment
  Tumour proliferation, indexed using Ki-67 immunohistochemistry, following treatment with neoadjuvant leuprolide, abiraterone acetate, and prednisone with and without cabazitaxel will be evaluated.
Androgen receptor expression | up to 24 weeks of treatment
  Androgen receptor expression will be evaluated using immunohistochemistry following treatment with neoadjuvant leuprolide, abiraterone acetate, and prednisone with and without cabazitaxel.
Incidence of adverse events | up to 24 weeks of treatment
  Incidence of adverse events will be evaluated for the duration of the study.
Severity of adverse events | Aup to 24 weeks of treatment
  Severity of adverse events will be evaluated for the duration of the study.
Androgen levels (if optional biopsy tissue is available) | up to 24 weeks of treatment
  If the participants agrees to optional pre-treatment biopsy, androgen levels will be compared between the pre-treatment tissue samples and prostatectomy tissue.
Genomic alterations between pre- and post-treatment tissue | up to 24 weeks of treatment
  If the participants agrees to optional pre-treatment biopsy, genomic alterations between the pre-treatment tissue samples and prostatectomy tissue will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Neil E Fleshner, MD, MPH, FRCSC, Principal Investigator — University Health Network, Toronto; Anthony Joshua, BSc (Med), MBBS, PhD, FRACP, Principal Investigator — University Health Network, Toronto
Locations (5):
- Canada (5):
  - The Prostate Centre, Vancouver, British Columbia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network, Princess Margaret Cancer Centre, Toronto, Ontario